CLINICAL TRIAL: NCT00231374
Title: In Vivo Analysis of Intradural Pressure Variation With Patient Positioning
Brief Title: Measure of Cerebrospinal Fluid (CSF) Pressure Variation With Patient Positioning
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting patients for the study.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, S. Tim Yoon, M.D., Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0489-2005
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Back Pain
Keywords: cerebrospinal fluid; pain in cervical spine; pain in lumbar spine; myelogram
MeSH Terms: conditions — Back Pain; Low Back Pain | interventions — Myelography

INTERVENTIONS:
Procedure: Myelogram

SUMMARY:
This is a study looking at pressure changes in the fluid that surrounds the spine when a person is positioned in 2-3 different ways.

DETAILED DESCRIPTION:
Volunteers who need a myelogram of their spine as part of their routine medical care are being asked to be in this study. A myelogram is an imaging study with x-rays after an agent is put into the spine that shows spinal fluid on the x-ray. It requires insertion of a needle into the cerebrospinal fluid (CSF) inside the spine. CSF is a bodily fluid that bathes the brain, spinal cord, and nerve roots. This study is being conducted to measure CSF pressure changes with different patient positioning.

We are motivated to do this research study to better treat patients who develop a spinal fluid leak during a myelogram or other spine procedure. The tissue that holds the cerebrospinal fluid (CSF) is called the dura. During surgery or other procedures, the dura can develop a tear. Dural tears can result in a leakage of CSF. CSF leaks are a recognized complication of spinal surgery. Currently, there is no evidence on whether or not a specific postoperative spine position is beneficial, especially for cervical (neck spine) CSF leaks. The process of dural healing after a dural tear is influenced by CSF pressure. High CSF pressure may inhibit dural healing. We want to find the patient position (sitting, lying down, or reclining) that reduces the CSF pressure the most. To do this, we want to attach a pressure monitor to the needle that is normally placed in the spine for a myelogram and measure the CSF pressure.

ELIGIBILITY:
Inclusion Criteria:

* Need a lumbar or cervical myelogram as part of routine care.

Exclusion Criteria:

* Not needing a myelogram in the cervical or lumbar spine.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
CSF pressure measurements on 5 patients having a cervical myelogram in 3 positions.
CSF pressure measurements on 5 patients having a lumbar myelogram in 2 positions.

SECONDARY OUTCOMES:
Safety measurements of one position over another.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Yoon, M.D., Principal Investigator — Emory University
Locations (1):
- Emory Orthopaedics & Spine Center, Atlanta, Georgia, United States

REFERENCES:
- See also: Departmental web site — http://www.emoryhealthcare.org/emory-orthopaedics-spine-hospital/index.html